CLINICAL TRIAL: NCT01607957
Title: Randomized, Double-blind, Phase 3 Study of TAS-102 Plus Best Supportive Care (BSC) Versus Placebo Plus BSC in Patients With Metastatic Colorectal Cancer Refractory to Standard Chemotherapies
Brief Title: Study of TAS-102 in Patients With Metastatic Colorectal Cancer Refractory to Standard Chemotherapies
Acronym: RECOURSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPU-TAS-102-301; 2012-000109-66 (EudraCT Number)
Record Dates: First submitted 2012-05-24; First posted 2012-05-30 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer
Keywords: Refractory, metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAS-102 (Experimental)
  Interventions: Drug: TAS-102
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAS-102 — 35 mg/m2/dose, orally, twice daily on days 1-5 and 8-12 of each 28-day cycle. Number of cycles: until at least one of the discontinuation criteria are met.
  Arms: TAS-102
Drug: Placebo — Placebo tablets, orally, twice daily on days 1-5 and 8-12 of each 28-day cycle. Number of cycles: until at least one of the discontinuation criteria are met.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the efficacy and safety of TAS-102 versus placebo in patients with refractory metastatic colorectal cancer.

DETAILED DESCRIPTION:
This is a multinational, double-blind, two-arm, parallel, randomized Phase 3 comparison study evaluating the efficacy and safety of TAS-102 versus placebo in patients with refractory metastatic colorectal cancer. Patients will be randomly assigned (2:1) to TAS-102 (experimental arm) or placebo (control arm).

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent
2. Has adenocarcinoma of the colon or rectum
3. Has failed at least 2 prior regimens of standard chemotherapies for metastatic colorectal cancer
4. ECOG performance status of 0 or 1
5. Is able to take medications orally
6. Has adequate organ function (bone marrow, kidney and liver)
7. Women of childbearing potential must have a negative pregnancy test and must agree to adequate birth control if conception is possible. Males must agree to adequate birth control.

Exclusion Criteria:

1. Certain serious illnesses or medical condition(s)
2. Has had certain other recent treatment e.g. major surgery, anticancer therapy, extended field radiation, received investigational agent, within the specified time frames prior to study drug administration
3. Has received TAS-102
4. Has unresolved toxicity of greater than or equal to CTCAE Grade 2 attributed to any prior therapies
5. Is a pregnant or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2012-06-17 (Actual); Primary Completion 2014-01-31 (Actual); Study Completion 2016-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: From - Boston, MA, Principal Investigator — Dana-Farber Cancer Institute; From - Leuven, Belgium, Principal Investigator — University Hospital, Gasthuisberg; From - Kashiwa, Chiba Japan, Principal Investigator — National Cancer Center Hospital East
Locations (114):
- United States (23):
  - Arizona Center for Cancer Care, Glendale, Arizona
  - California Cancer Associates for Research and Excellence, Fresno, California
  - Ronald H. Yanagihara, MD, Gilroy, California
  - LAC and USC Medical Center, Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - San Jose Medical Group, San Jose, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Yale Cancer Center, New Haven, Connecticut
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Illinois Cancer Care, P.C., Peoria, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Clinic Fndtn, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Jefferson City Medical Group, Jefferson City, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Gabrail Cancer Center, Canton, Ohio
  - Hickman Cancer Center at Flower Hospital, Sylvania, Ohio
  - Hematology/Oncology Associates of Fredericksburg, Fredericksburg, Virginia
- Australia (5):
  - Royal North Shore Hospital, Sydney, New South Wales
  - The Queen Elisabeth Hospital, Woodville South, South Australia
  - Austin Hospital, Heidelberg, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- Austria (5):
  - Krankenhaus der Barmherzigen Schwestern Linz, Linz
  - Universitaet Wien, Vienna
  - Universitaetsklinik fur Innere Medizin, Vienna
  - Wilhelminenspital Wien, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Belgium (8):
  - Cliniques Universitaires UCL St. Luc, Brussels
  - Erasme University Hospital-ULB-Brussels, Brussels
  - Grand Hospital de Charleroi, Charleroi
  - Antwerp University Hospital, Edegem
  - University Hospital Gent, Edegem
  - University Hospital Gent, Ghent
  - Leuven University Hospital - Campus Gasthuiseberg, Leuven
  - University Hospital Gasthuisberg, Leuven
- Czechia (2):
  - Klinika onkologie a radioteraie, Facultni nemocnice Hradec Kralove, Hradec Králové
  - Institute of Oncology and Rehabilitation Ples, Nová Ves pod Pleší
- France (6):
  - CHU de Becançon, Besançon
  - University Hospital of Bordeaux, Bordeaux
  - Centre Oscar Lambret, Lille
  - CRLC Val d'Aurelle, Montpellier
  - Hopital Saint Antoine, Paris
  - Centre Eugene Marquis, Rennes
- Germany (13):
  - Onkologische Schwerpunktpraxis Kurfuerstendamm, Berlin
  - Praxiskooperation Bonn-Euskirchen-Rheinbach, Bonn
  - Uniklinik Koeln, Cologne
  - Universitatsklinikum Carl Gustav Carus - Dresden, Dresden
  - Medizinische Klinik am Krankenhaus Nordwest GmbH, Frankfurt
  - Uniklinik der Martin-Luther-Universitaet Halle-Wittenberg, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Johannes Gutenberg Universität Mainz, Mainz
  - Interdisziplinaeres Tumorzentrum Mannheim, Mannheim
  - Klinikum der Universität München - Großhadern, München
  - Staedtisches Klinikum Muenchen / Klinikum Neuperlach, München
  - Klinikum Oldenburg gGmbH, Oldenburg
  - Universitaetsklinikum Ulm, Ulm
- Ireland (3):
  - Bon Secours Hospital, Cork
  - Adelaide and Meath Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
- Italy (11):
  - Fondazione Poliambulanza, Brescia, Lombardy
  - Universita Delgi Studi de Genova (UNIGE)- Azienda Ospedaliera. Universitaria "San Martino" (Ospedale San Martino), Genova
  - A.O. Ospedale Niguarda Ca' Granda, Milan
  - Fondazione IRCCS Instituto Nazionale dei Tumori Milano, Milan
  - A.O. R.N. "A.Cardarelli", Naples
  - Seconda Universita degli Studi de Napoli, Napoli
  - AOU San Luidi di Orbassano, Orbassano
  - Azienda Ospedaliero, Pisa
  - Arcispidale S Maria Nuova, Reggio Emilia
  - Ospedale di Rimini, Rimini
  - Ospedale di Sondrio, Sondrio
- Japan (20):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - KKR Sapporo Medical Center TONAN-Hospital, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Tsukuba University Hospital, Tsukuba, Ibaraki
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Osaka Medical College Hospital, Takatsuki, Osaka
  - Saitama Cancer Center, Kita-adachi-gun, Saitama
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Chiba Cancer Center, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kumamoto University Hospital, Kumamoto
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka
  - Tokushima University Hospital, Tokushima
- Spain (11):
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital Arnau de Vilanova, Lleida
  - Hospital Universitario Ramon y Cajal, Madrid
  - Fundacion Jimenez Diaz - Universidad Autonoma de Madrid, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Carlos Haya, Málaga
  - Hospital Universitario Morales Messeguer, Murcia
  - Corporacion Sanitaria Parc Tauli, Sabadell
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Akademiska Sjukhuset, Uppsala
- United Kingdom (5):
  - Aberdeen Royal Infirmary, Aberdeen
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - St James' Institute of Oncology, Leeds
  - University College London Hospitals Foundation NHS Trust, London
  - The Royal Marsden NHS Foundation Trust, Surrey

REFERENCES:
- [Derived] Yoshino T, Cleary JM, Van Cutsem E, Mayer RJ, Ohtsu A, Shinozaki E, Falcone A, Yamazaki K, Nishina T, Garcia-Carbonero R, Komatsu Y, Baba H, Argiles G, Tsuji A, Sobrero A, Yamaguchi K, Peeters M, Muro K, Zaniboni A, Sugimoto N, Shimada Y, Tsuji Y, Hochster HS, Moriwaki T, Tran B, Esaki T, Hamada C, Tanase T, Benedetti F, Makris L, Yamashita F, Lenz HJ. Neutropenia and survival outcomes in metastatic colorectal cancer patients treated with trifluridine/tipiracil in the RECOURSE and J003 trials. Ann Oncol. 2020 Jan;31(1):88-95. doi: 10.1016/j.annonc.2019.10.005. PMID 31912801
- [Derived] Van Cutsem E, Mayer RJ, Laurent S, Winkler R, Gravalos C, Benavides M, Longo-Munoz F, Portales F, Ciardiello F, Siena S, Yamaguchi K, Muro K, Denda T, Tsuji Y, Makris L, Loehrer P, Lenz HJ, Ohtsu A; RECOURSE Study Group. The subgroups of the phase III RECOURSE trial of trifluridine/tipiracil (TAS-102) versus placebo with best supportive care in patients with metastatic colorectal cancer. Eur J Cancer. 2018 Feb;90:63-72. doi: 10.1016/j.ejca.2017.10.009. Epub 2017 Dec 21. PMID 29274618
- [Derived] Longo-Munoz F, Argiles G, Tabernero J, Cervantes A, Gravalos C, Pericay C, Gil-Calle S, Mizuguchi H, Carrato-Mena A, Limon ML, Garcia-Carbonero R. Efficacy of trifluridine and tipiracil (TAS-102) versus placebo, with supportive care, in a randomized, controlled trial of patients with metastatic colorectal cancer from Spain: results of a subgroup analysis of the phase 3 RECOURSE trial. Clin Transl Oncol. 2017 Feb;19(2):227-235. doi: 10.1007/s12094-016-1528-7. Epub 2016 Jul 21. PMID 27443414
- [Derived] Mayer RJ, Van Cutsem E, Falcone A, Yoshino T, Garcia-Carbonero R, Mizunuma N, Yamazaki K, Shimada Y, Tabernero J, Komatsu Y, Sobrero A, Boucher E, Peeters M, Tran B, Lenz HJ, Zaniboni A, Hochster H, Cleary JM, Prenen H, Benedetti F, Mizuguchi H, Makris L, Ito M, Ohtsu A; RECOURSE Study Group. Randomized trial of TAS-102 for refractory metastatic colorectal cancer. N Engl J Med. 2015 May 14;372(20):1909-19. doi: 10.1056/NEJMoa1414325. PMID 25970050

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted in 101 study centers in 13 countries including the United States, Japan, Spain, Italy, Germany, Belgium, France, Australia, United Kingdom, Austria, Ireland, Sweden, and Czech Republic.
Pre-assignment Details: Total 1002 participants provided consent, out of which 800 participants were randomized in 2:1 ratio in TAS-102 and placebo treatment groups respectively.
Groups:
- TAS-102: Participants received TAS-102 orally with a starting dose of 35 milligram per meter square per dose (mg/m^2/dose) twice daily (BID) based on body surface area (BSA) along with best supportive care (BSC). The first dose of TAS-102 was administered in the morning of Day 1 of each cycle and the last dose was administered in the evening of Day 5, followed by rest on Day 6 and 7. The treatment was repeated for next week starting from Day 8 to Day 12, followed by a 16-day rest starting from Day 13 to Day 28 (1 treatment cycle = 28 days). Participants received study medication until any of the discontinuation criteria were met.
- Placebo: Participants orally received TAS-102 matching placebo BID dose along with BSC with the first dose administered in the morning of Day 1 of each cycle and the last dose administered in the evening of Day 5, followed by rest on Day 6 and 7. The treatment was repeated for next week starting from Day 8 to Day 12, followed by a 16-day rest starting from Day 13 to Day 28 (1 treatment cycle). Participants received study medication until any of the discontinuation criteria.
Period: Overall Study
Arm/Group | TAS-102 | Placebo
Started | 534 | 266
Treated | 533 | 265
Completed | 162 | 51
Not Completed | 372 | 215
Not completed — Not treated | 1 | 1
Not completed — Death | 367 | 211
Not completed — Lost to Follow-up | 3 | 3
Not completed — Participant refusal | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed in Intent-to-Treat (ITT) population which included all randomized participants.
Groups:
- TAS-102: Participants received TAS-102 orally with a starting dose of 35 mg/m^2/dose BID based on BSA along with BSC. The first dose of TAS-102 was administered in the morning of Day 1 of each cycle and the last dose was administered in the evening of Day 5, followed by rest on Day 6 and 7, treatment was repeated for next week starting from Day 8 to Day 12, followed by a 16-day rest starting from Day 13 to Day 28 (1 treatment cycle = 28 days). Participants received study medication until any of the discontinuation criteria were met.
- Placebo: Participants orally received TAS-102 matching placebo BID dose along with BSC with the first dose administered in the morning of Day 1 of each cycle and the last dose administered in the evening of Day 5, followed by rest on Day 6 and 7, treatment was repeated for next week starting from Day 8 to Day 12, followed by a 16-day rest starting from Day 13 to Day 28 (1 treatment cycle). Participants received study medication until any of the discontinuation criteria.
- Total: Total of all reporting groups
Arm/Group | TAS-102 | Placebo | Total
Number analyzed (Participants) | 534 | 266 | 800
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 300 | 148 | 448
  >=65 years | 234 | 118 | 352
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (10.21) | 61.5 (10.51) | 61.5 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 208 | 101 | 309
  Male | 326 | 165 | 491

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of randomization to the date of death for participants. If a participant discontinued study medication for reasons other than radiologic disease progression, the participant was followed for tumor response until radiologic disease progression or initiation of new anticancer therapy.
Time Frame: Every 8 weeks, up to 12 months after the last participant was randomized or until the target number of events (deaths) was met, whichever was later. (Overall survival data was collected till 24 Jan 2014 which was date of observation of the 571st death)
Population: Analysis was performed in ITT population. For participants who were alive as of the overall survival cutoff date, their survival was censored on the cutoff date post consent.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TAS-102 | Placebo
Number analyzed (Participants) | 534 | 266
months | 7.1 [6.5 to 7.8] | 5.3 [4.6 to 6.0]
Statistical Analysis 1: Comparison: TAS-102 vs Placebo; Test type: Superiority; p < 0.0001, Stratified log-rank test; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.58 to 0.81]

2. Secondary Outcome: Progression-free Survival
Description: Tumor assessments were performed throughout the study based on RECIST, Version 1.1, 2009. Progression free survival was defined as the time (in months) from the date of randomization until the date of the investigator-assessed radiological disease progression or death due to any cause. For participants who were alive with no radiological disease progression as of the analysis cut-off date, their survival was censored at the date of the last tumor assessment. Participants who received non-study cancer treatment before disease progression, or participants with clinical but not radiologic evidence of progression, were censored at the date of the last radiologic evaluable tumor assessment before the non-study cancer treatment was initiated.
Time Frame: Every 8 weeks, up to 12 months after the last participant was randomized or until the date of the investigator-assessed radiological disease progression or death due to any cause,whichever was later. (Progression free survival cutoff: 31 Jan 2014)
Population: Analysis was performed in ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TAS-102 | Placebo
Number analyzed (Participants) | 534 | 266
months | 2.0 [1.9 to 2.1] | 1.7 [1.7 to 1.8]
Statistical Analysis 1: Comparison: TAS-102 vs Placebo; Test type: Superiority; p < 0.0001, Stratified log-rank test; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.41 to 0.57]

3. Secondary Outcome: Percentage of Participants With Adverse Events (AE), Treatment-Related AEs, Discontinuations, Serious Adverse Events (SAEs) and Deaths
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-related AEs were events between administration of study drug and up to 30 Days that were absent before treatment or that worsened relative to pre-treatment state. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability /incapacity; congenital anomaly. The AEs were graded for severity using National Cancer Institute Common Terminology Criteria for AEs.
Time Frame: From the time of signing the informed consent form until the period of participant follow up (30 days following after the administration of last dose of study medication or until initiation of new antitumor therapy, whichever was earlier
Population: Safety analysis was performed on as treated (AT) population including all participants who took part of any dose of the study medication.
Measure: Number; unit: percentage of participants
Arm/Group | TAS-102 | Placebo
Number analyzed (Participants) | 533 | 265
percentage of participants
  Any adverse event (AE) | 98.3 | 93.2
  Any treatment-related AE | 85.7 | 54.7
  Any ≥Grade 3 AE | 69.4 | 51.7
  Any treatment-related ≥Grade 3 AE | 49.0 | 9.8
  Any serious AE (SAE) | 29.6 | 33.6
  Any AE resulting in discontinuation | 10.3 | 13.6
  Any AE with outcome of death | 3.2 | 11.3

ADVERSE EVENTS:
Time Frame: From the time of signing the informed consent form until the period of participant follow up (30 days following the administration of last dose of study medication or until initiation of new anti-tumor therapy, whichever was earlier, up to 85 weeks approximately (duration of study)).
Description: Safety analysis was performed on AT population including all participants who took part of any dose of the study medication.
Arm/Group | TAS-102 | Placebo
All-Cause Mortality (participants affected / at risk) | 17/533 | 30/265
Serious Adverse Events (participants affected / at risk) | 158/533 | 89/265
Other Adverse Events (participants affected / at risk) | 506/533 | 227/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAS-102 (N=533) | Placebo (N=265)
Anaemia (Blood and lymphatic system disorders) | 10 (10) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 14 (14) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-Respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 5 (5)
Ascites (Gastrointestinal disorders) | 3 (3) | 3 (3)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 3 (3) | 5 (5)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sigmoiditis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 5 (6) | 1 (3)
Subileus (Gastrointestinal disorders) | 2 (3) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (7) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (3) | 2 (2)
General physical health deterioration (General disorders) | 15 (15) | 11 (11)
Hyperpyrexia (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Multi-Organ failure (General disorders) | 1 (1) | 0 (0)
Obstruction (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (5) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 3 (3) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 3 (3) | 6 (6)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 3 (3) | 2 (2)
Jaundice cholestatic (Hepatobiliary disorders) | 4 (4) | 2 (2)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Biliary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (4)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Brain compression (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 2 (2) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2) | 1 (1)
Epiduritis (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1)
Nerve root compression (Nervous system disorders) | 1 (1) | 0 (0)
Neurological decompensation (Nervous system disorders) | 0 (0) | 1 (1)
Psychomotor skills impaired (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Postrenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 5 (5) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Intra-Abdominal haematoma (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAS-102 (N=533) | Placebo (N=265)
Anaemia (Blood and lymphatic system disorders) | 205 (265) | 22 (24)
Leukopenia (Blood and lymphatic system disorders) | 27 (34) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 152 (327) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 35 (58) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 74 (83) | 32 (32)
Abdominal pain upper (Gastrointestinal disorders) | 38 (40) | 12 (15)
Constipation (Gastrointestinal disorders) | 81 (87) | 40 (42)
Diarrhoea (Gastrointestinal disorders) | 167 (240) | 33 (39)
Nausea (Gastrointestinal disorders) | 256 (410) | 63 (73)
Stomatitis (Gastrointestinal disorders) | 42 (54) | 16 (17)
Vomiting (Gastrointestinal disorders) | 142 (217) | 38 (57)
Asthenia (General disorders) | 96 (116) | 29 (29)
Fatigue (General disorders) | 185 (227) | 60 (64)
Mucosal inflammation (General disorders) | 30 (37) | 12 (13)
Oedema peripheral (General disorders) | 52 (57) | 27 (27)
Pyrexia (General disorders) | 93 (115) | 36 (40)
Alanine aminotransferase increased (Investigations) | 25 (31) | 14 (14)
Aspartate aminotransferase increased (Investigations) | 30 (33) | 21 (22)
Blood alkaline phosphatase increased (Investigations) | 47 (48) | 26 (26)
Blood bilirubin increased (Investigations) | 44 (59) | 18 (19)
Neutrophil count decreased (Investigations) | 148 (417) | 1 (12)
Platelet count decreased (Investigations) | 81 (172) | 6 (6)
Weight decreased (Investigations) | 40 (44) | 27 (27)
White blood cell count decreased (Investigations) | 146 (354) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 206 (276) | 76 (81)
Hyponatraemia (Metabolism and nutrition disorders) | 15 (16) | 14 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 39 (41) | 18 (18)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 28 (30) | 20 (21)
Dysgeusia (Nervous system disorders) | 36 (42) | 6 (6)
Headache (Nervous system disorders) | 29 (32) | 13 (14)
Insomnia (Psychiatric disorders) | 24 (24) | 25 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 56 (61) | 30 (32)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 54 (59) | 28 (28)
Alopecia (Skin and subcutaneous tissue disorders) | 36 (36) | 3 (3)
Hypertension (Vascular disorders) | 19 (23) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Taiho agreements vary with individual investigators, but do not prohibit any from publishing. Taiho is provided time to review material discussing trial results (generally 30 to 120 days with possible extension), and can remove undisclosed confidential, proprietary and intellectual property rights-related information. Authors have final control and approval of publication content of final study results. The investigator agrees not to publish any results before the first multicenter publication.